CLINICAL TRIAL: NCT02376660
Title: A Randomized Controlled Trial to Evaluate the Efficacy of 3 g of Soluble Fiber From Oats on the Lipid Profile of Men and Women With Elevated Lipid Levels Aged Between 20 and 50 Years
Brief Title: Effect of Oats on Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1205
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Mildly Hypercholesterolemic Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oats (Experimental): 70 grams oats
  Interventions: Other: Oats
- usual diet and exercise (Placebo Comparator): usual diet and exercise

INTERVENTIONS:
Other: Oats
  Arms: Oats

SUMMARY:
A randomized control trial to assess the effect of oats on lipid profile of mildly hypercholesterolemic subjects. Subjects consumed 35g of oats twice daily (total of 70g / day) in place of carbohydrates as part of their usual diet. 70 grams of oats provide 3 grams of soluble fiber. Control group consumed the usual diet. Subjects followed up for 4 weeks. In total 3 assessment visits of the subjects planned for the study period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 50 years old
* Total Cholesterol: ≥ 200 mg/dL and < 240mg/dL
* Availability and willingness to follow study protocol
* Stable body weight for previous 3 months (not more than 5% weight change)

Exclusion Criteria:

* Subjects already on lipid lowering drugs
* LDL-c > 190 mg/dL
* Total cholesterol <200 mg/dL and >240 mg/dL
* Subjects with serum creatinine levels > 1.3 mg/dL (female) or 1.4 mg/dL (male), nephropathy, evidence of hepatic disease or history of alcohol abuse
* Baseline Triglycerides: > 300 mg/dL
* Diabetes (Type 1 or Type 2) as diagnosed by a physician
* Uncontrolled hyperthyroidism (as per physician's discretion)
* Uncontrolled hypertension (as per physician's discretion)
* Acute infections or chronic debilitating diseases like tuberculosis, malignancy, HIV infection etc. Any life threatening serious disorder of the liver, kidneys, heart, lungs or other organs by history
* Irritable bowel syndrome by history
* Unwillingness to give written informed consent for participation in the study.
* Pregnancy & lactation (by history)
* Severe end organ damage
* Subjects with allergy to oats
* Heavy smokers (smoking more than 5 cigarettes per day)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
reduction of total cholesterol | 4 weeks

SECONDARY OUTCOMES:
LDL-c | 4 weeks
Triglycerides | 4 weeks
Blood pressure | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, MBBS, Principal Investigator — Fortis Clinical Research Limited

REFERENCES:
- [Derived] Gulati S, Misra A, Pandey RM. Effects of 3 g of soluble fiber from oats on lipid levels of Asian Indians - a randomized controlled, parallel arm study. Lipids Health Dis. 2017 Apr 4;16(1):71. doi: 10.1186/s12944-017-0460-3. PMID 28376899